CLINICAL TRIAL: NCT06903273
Title: Neoadjuvant Tislelizumab, Gemcitabine, Cisplatin and S-1 for Patients with Resectable High-risk Intrahepatic Cholangiocarcinoma
Brief Title: Neoadjuvant Tislelizumab, Gemcitabine, Cisplatin and S-1 for Resectable High-risk Cholangiocarcinoma
Acronym: TisGCS for BTC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Kaohsiung Veterans General Hospital. (Other); Chi Mei Medical Hospital (Other)
Responsible Party: Principal Investigator, Chih Chieh, Yen, Principal Investigator, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCKUH-BTC-01
Record Dates: First submitted 2025-03-18; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cholangiocarcinoma; Biliary Tract Cancer (BTC)
Keywords: cholangiocarcinoma; biliary tract cancer; neoadjuvant; gemcitabine; S-1; preoperative; resectable; tislelizumab; cisplatin
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms | interventions — tislelizumab; Gemcitabine; Cisplatin; S 1 (combination)

STUDY DESIGN:
Intervention Model Description: Simon two-staged design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab-Gemcitabine/Cisplatin/S-1 (Experimental): neoadjuvant tislelizumab/gemcitabine/cisplatin/S-1
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab plus chemotherapy (14 days as one cycle) 3 cycles every 2 weeks as neoadjuvant therapy and followed by a curative surgery.
  Tislelizumab 200 mg fixed-dose IVD on day 1. Gemcitabine 800 mg/m2 on day 1 with a fixed-infusion rate of 80 mins. Cisplatin 25 mg/m2 on day 1. S-1 70 mg/m2 daily as a BID dosing per oral on day 1 to 7. (daily total dose determined by body surface area (BSA): <1.25 m2, 80 mg; 1.25-1.50 m2, 100 mg; ≥1.50 m2, 120 mg)
  Other Names: gemcitabine; cisplatin; S-1

SUMMARY:
To investigate the efficacy and tolerability of neoadjuvant tislelizumab, gemcitabine, cisplatin and S-1 (TisGCS) in patients with resectable high-risk iCCA.

DETAILED DESCRIPTION:
Patients with cholangiocarcinoma have limited therapeutic options and a poor prognosis. Margin-free resection is the only curative treatment to treat intrahepatic cholangiocarcinoma (iCCA). However, patients with resectable disease still suffer from high recurrence or progression. Both immune checkpoint inhibitors and chemotherapy have shed light on treating patients with iCCA. Nevertheless, the role of neoadjuvant chemo-immunotherapy has not been established in patients with resectable iCCA harboring a high risk for recurrence. The aim of the trial is to investigate the efficacy and tolerability of neoadjuvant tislelizumab, gemcitabine, cisplatin and S-1 (Tis-GCS) in patients with resectable high-risk iCCA. The primary outcome is R0 resection rate. The secondary outcome includes objective response rate, event-free survival, overall survival, protocol completion rate and adverse events. The study is an open-label, single-arm and multi-center phase II investigator-initiated trial with Simon two-stage design. Subjects with resectable iCCA harboring a high risk for recurrence or those suffer from very early recurrent disease who are eligible for a curative resection are included. A total of 35 subjects are expected with a minimal sample size of 14 when the R0 resection rate is of the lower threshold. Tis-GCS (14 days as a cycle) 3 cycles every 2 weeks will be administered and followed by surgery. Tislelizumab 200 mg fixed-dose, gemcitabine 800 mg/m2 and cisplatin 25 mg/m2 is given intravenously on day 1. S-1 (35 mg/m2) is given twice daily per oral on day 1 to 7. The study will prove the feasibility and efficacy of neoadjuvant chemo-immunotherapy in resectable high-risk iCCA. The results may provide critical fundamentals into future phase III clinical trials.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must meet the criteria of either (A) or (B), plus 1. to 6. (A) High-risk group (HR) Subjects have histologically-confirmed and potentially resectable intrahepatic cholangiocarcinoma, according to the definition of American Joint Cancer Committee staging system, 8th edition (AJCC 8th).

Plus at least one of the following high-risk features,

1. Solitary tumor with a maximal diameter ≥5 cm in the absence of vascular invasion.
2. ≥T1b disease which is resectable.
3. Multifocal tumors or single tumor with satellite nodules at the same anatomic liver lobe which is/are resectable.
4. Tumor(s) with macroscopic intrahepatic vascular invasion but is/are potentially resectable.
5. Image or histological evidence of hilar or portal lymph node involvement (N1).
6. Initial serum cancer antigen-199 (CA199) ≥200 U/mL.

   (B) Very early recurrence group (VER) Subjects with previously resected cholangiocarcinoma under a curative intent and have an early recurrent disease (≤6 months post curative surgery) confined to the liver, with/without antecedent adjuvant local or systemic therapies, and can be re-resected under a curative intent.
   1. Subjects present with at least one measurable lesion which can be accurately assessed by conventional techniques at least 1.0 cm by computed tomography (CT) or magnetic resonance imaging (MRI).
   2. Subjects are above 18 years of age with an Eastern Cooperative Oncology Group (ECOG) performance status ≤1, have a life expectancy >3 months, have surgically resectable disease and are physically competent and willing to receive a curative operation following the study protocol
   3. Subjects have adequate organ functions, including bone marrow reserve with a leukocyte count ≥3,000 /µL and platelet count ≥50,000 /µL, hepatic reserve with a serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) and total bilirubin ≤3 times of upper normal testing limits (biliary drainage is permitted), renal reserve with a creatinine clearance ≥60 mL/min and cardiac reserve with a New York Heart Association (NYHA) functional classification I at baseline.
   4. Subjects have or agree to establish a vascular access that permits intravenous administration of medications and are capable of ingesting capsules per oral.
   5. Subjects with reproductive potentials are willing to accept contraceptive measures during the trial.
   6. Subjects are functionally and cognitively capable to be informed of the trial contents and objectives (including obtaining blood and tumor tissue for the trial investigation), and agree to sign the written consent for enrollment.

   Exclusion Criteria:
   1. Subjects have metastatic (M1) disease, recurrent cholangiocarcinoma which cannot be resected, recurrent cholangiocarcinoma which can be re-resected but occurs >6 months post previous surgery, or any other primary malignancies in which the subjects have been in disease-free status less than 2 years, excluding carcinoma in situ or resectable skin cancer.
   2. Subjects have received a systemic therapy with either chemotherapeutics or immune checkpoint inhibitors, a major abdominal surgery or radiotherapy within 4 weeks before the trial enrollment.
   3. Subjects are known to be severely allergic to any of the studied therapeutics.
   4. Subjects have underlying chronic illnesses, including cardiopulmonary diseases, ischemic heart disease, inflammatory bowel disease, poorly-controlled diabetes mellitus, liver cirrhosis and/or debilitating autoimmune diseases or conditions.

   5 Subjects are receiving or have received a systemic administration of an equivalent dose of daily 10 mg prednisone or above for ≥14 days in whatever indications within 4 weeks before the trial enrollment, or immunosuppressives for ≥7 days within 4 weeks before the trial enrollment.

   6. Subjects have active bacterial, viral, fungal or mycobacterial infections that require systemic therapy, including active infection with human immunodeficiency virus (HIV), hepatitis B or C virus (HBV or HCV).

   7. Subjects are planning to conceive or already in pregnancy or breastfeeding. 8. Subjects are currently participating in any other clinical trials or studies which potentially interfere the protocol commencement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | From enrollment to surgical resection at 2 weeks
  Margin-free resection (R0) rate: (Number of patients with surgical results achieving an uninvolved margin under microscopic and macroscopic inspection) / (Number of patients receiving a surgery) x 100%

SECONDARY OUTCOMES:
Objective response rate | From enrollment to the end of neoadjuvant therapy at 2 weeks
  Patients who achieve a complete or partial response as defined by revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Overall survival | From the date of enrollment until the date of death from any cause
  The time interval from enrollment to death by any causes
Event-free survival | From the date of enrollment until the date of any predefined event which happens first
  The time interval from enrollment to an event, defined as disease progression, recurrence, withdrawal from trial treatment, initiation of subsequent anticancer treatment or death by any cause, in whichever happens first.
Disease control rate | From enrollment to the end of neoadjuvant therapy at 2 weeks
  Patients who achieve a complete response, partial response or stable disease, as defined by revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

OTHER OUTCOMES:
Protocol completion rate | From enrollment to the end of neoadjuvant therapy at 2 weeks
  Patients who complete the protocol neoadjuvant treatment / Enrolled patients X100%
Adverse events related to protocol treatment | From enrollment to the end of neoadjuvant therapy at 2 weeks
  Patients who present with ≥grade III adverse events resulting from protocol treatment per National Cancer Institute- Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Chia Jui Yen, MD., PhD, Principal Investigator — Department on Oncology, National Cheng Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol, SAP
Time Frame: 01/Jul/2025 to 01/Jul/2028
Access Criteria: Reviewers with a reasonable request to the principal investigator, Dr. Chih Jui, YEN.

REFERENCES:
- [Background] Maithel SK, Keilson JM, Cao HST, Rupji M, Mahipal A, Lin BS, Javle MM, Cleary SP, Akce M, Switchenko JM, Rocha FG. NEO-GAP: A Single-Arm, Phase II Feasibility Trial of Neoadjuvant Gemcitabine, Cisplatin, and Nab-Paclitaxel for Resectable, High-Risk Intrahepatic Cholangiocarcinoma. Ann Surg Oncol. 2023 Oct;30(11):6558-6566. doi: 10.1245/s10434-023-13809-5. Epub 2023 Jun 27. PMID 37368098
- [Background] Oh DY, Ruth He A, Qin S, Chen LT, Okusaka T, Vogel A, Kim JW, Suksombooncharoen T, Ah Lee M, Kitano M, Burris H, Bouattour M, Tanasanvimon S, McNamara MG, Zaucha R, Avallone A, Tan B, Cundom J, Lee CK, Takahashi H, Ikeda M, Chen JS, Wang J, Makowsky M, Rokutanda N, He P, Kurland JF, Cohen G, Valle JW. Durvalumab plus Gemcitabine and Cisplatin in Advanced Biliary Tract Cancer. NEJM Evid. 2022 Aug;1(8):EVIDoa2200015. doi: 10.1056/EVIDoa2200015. Epub 2022 Jun 1. PMID 38319896
- [Background] Kelley RK, Ueno M, Yoo C, Finn RS, Furuse J, Ren Z, Yau T, Klumpen HJ, Chan SL, Ozaka M, Verslype C, Bouattour M, Park JO, Barajas O, Pelzer U, Valle JW, Yu L, Malhotra U, Siegel AB, Edeline J, Vogel A; KEYNOTE-966 Investigators. Pembrolizumab in combination with gemcitabine and cisplatin compared with gemcitabine and cisplatin alone for patients with advanced biliary tract cancer (KEYNOTE-966): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 3;401(10391):1853-1865. doi: 10.1016/S0140-6736(23)00727-4. Epub 2023 Apr 16. PMID 37075781
- [Background] Ioka T, Kanai M, Kobayashi S, Sakai D, Eguchi H, Baba H, Seo S, Taketomi A, Takayama T, Yamaue H, Takahashi M, Sho M, Kamei K, Fujimoto J, Toyoda M, Shimizu J, Goto T, Shindo Y, Yoshimura K, Hatano E, Nagano H; Kansai Hepatobiliary Oncology Group (KHBO). Randomized phase III study of gemcitabine, cisplatin plus S-1 versus gemcitabine, cisplatin for advanced biliary tract cancer (KHBO1401- MITSUBA). J Hepatobiliary Pancreat Sci. 2023 Jan;30(1):102-110. doi: 10.1002/jhbp.1219. Epub 2022 Aug 9. PMID 35900311